CLINICAL TRIAL: NCT01484535
Title: Aspiration for Pain Relief Following Ankle Fracture: A Prospective Double-Blind Randomized Controlled Trial
Brief Title: Aspiration for Pain Relief Following Ankle Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen A. Sems, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 11-004187
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Ankle Fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ankle aspiration (Other): ankle aspiration
  Interventions: Procedure: Ankle Aspiration
- placebo procedure (Placebo Comparator): placebo procedure
  Interventions: Procedure: Ankle aspiration Standard Anterolateral

INTERVENTIONS:
Procedure: Ankle Aspiration — Ankle aspiration will be performed through either a standard anterolateral or anteromedial approach, depending on the conditions of the soft tissue. The anterolateral approach will be the preferred method due to the higher reproducibility of intra-articular needle placement. The anteromedial approach will be reserved for patients whose soft tissues over the anterolateral portal are compromised. Sterile preparation of the limb will be achieved with the use of chlorhexidine or Betadine. An 18 gauge needle will be introduced into the ankle joint and a syringe will be used to aspirate the ankle until no more hemarthrosis is able to be removed. The amount of hemarthrosis aspirated will be recorded. Following the procedure, care will continue as per standard of care.
  Arms: Ankle aspiration
Procedure: Ankle aspiration Standard Anterolateral — Placebo ankle aspiration will be performed through a standard anterolateral. Sterile preparation of the limb will be achieved with the use of chlorhexidine or Betadine. An 18-gauge needle will be introduced into the skin. The needle will be held in the skin for 5-10 seconds in an effort to simulate the pain and time-lag experienced with aspiration. The needle will not pass the fascia or ankle joint capsule. Following the procedure, care will continue as per standard of care.
  Arms: placebo procedure

SUMMARY:
This trial will study the effect of hematoma aspiration in patients with acute ankle fractures.

ELIGIBILITY:
Inclusion criteria:

* AO/OTA fracture classification 44
* Closed fracture
* Injury within 24 hours of presentation
* Skeletally mature
* Able to provide consent to participate in study

Exclusion Criteria:

* Any concomitant injuries affecting Numerical Rating Scale
* Soft tissue wounds at aspiration sites that compromise ability to aspirate
* Patient not able to complete pain medication log
* Patient not able to participate in follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain as rated by numerical rating scale (NRS) scores in the emergency department and in the first 72 hours from the time of initial evaluation. | 6 months
  Total amount of pain medication used in the first 72 hours from time of initial evaluation.

SECONDARY OUTCOMES:
Percentage of volumetric increase of the injured ankle compared to the uninjured ankle. | 6 months
  NRS scores after 72 hours through 6 months. 6 month SMFA scores. 6 month Olerud Molander scores.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Sems, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States